CLINICAL TRIAL: NCT00454311
Title: Prospective and Randomized Study of the Impact of the Biopsy of 1-2 Cells in a PGD Program for Aneuploidy Screening
Brief Title: The Impact of the Biopsy of 1-2 Cells in a PGD Program for Anueploidy Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Carmen Rubio, IVI Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: VLC-CR-1106-307-5
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Pregnancy and implantation rates; Efficiency and accuracy of the genetic testing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- One cell biopsy (Active Comparator)
  Interventions: Procedure: · day embryo biopsy
- Two cell biopsy (Other)
  Interventions: Procedure: Biopsy of Day 3 Embryo

INTERVENTIONS:
Procedure: Biopsy of Day 3 Embryo
  Arms: Two cell biopsy
Procedure: · day embryo biopsy
  Arms: One cell biopsy

SUMMARY:
The aim of this study is to evaluate the impact of the biopsy of one or two cells in a preimplantatation genetic diagnosis program (PGD) for the screening of aneuploidies. This prospective and randomized study will be performed at the Instituto Valenciano de Infertilidad in Valencia (Spain) in those patientes included in our clinical program. Our purpose is to optimize the methodology employed in our laboratory in order to guarantee optimal implantation and pregnancy rates without a detrimental effect on the accuracy and efficiency of the cytogenetic analysis. Patients will undergo and IVF cycle, embryo biopsy will be performed on day 3 embryos in two fashions: in some patients only one cell per embryo will be retrieved whereas in others, 2 cells will be retrieved in good morphology embryos and only 1 in the slowl ones. In all cases aneuploidy screening will be performed by FISH for chromosomes 13, 16, 18, 21, 22, X and Y. Embryo developmente will be checked every 24 hours and chormosomally normal embryos will be replaced into the uterus on day 5 of development.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PGD for aneuploidy screening with their own oocytes and for chromosomes 13, 16, 18, 21, 22, X & Y

Exclusion Criteria:

* Patients undergoing PGD for monogenic diseases (PCR)
* Patients undergoing PGD for structural chromosomal abnormalities
* Ovum donation cycles
* Cryopreserved oocyte/embryos

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
impact of biopsy | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Rubio, PhD, Principal Investigator — Instituto Valenciano de Infertilidad
Locations (1):
- Instituto Valenciano de la Infertilidad, Valencia, Spain